CLINICAL TRIAL: NCT04933136
Title: A Prospective Registry for the Evaluation of the Safety, Efficacy and Clinical Impact of the Double Hemostasis System Terry2 (TM) on Patients Undergoing a Trans-radial or Trans-cubital Catheterism.
Brief Title: Radial Artery Occlusion and Dual Artery Hemostasis After Transradial Approach.
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Tomas Cieza Lara, Principal Investigator, Laval University
Other Study IDs: Registry-Terry2 Band
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Radial Artery Occlusion
Keywords: Radial Artery Occlusion; Transradial approach; Transulnar approach; Dual artery hemostasis; Patent hemostasis
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Terry2 Band — Hemostasis protocol following radial or cubital approach catheterization using the dual artery hemostasis device Terry2Band.

SUMMARY:
* Improving patient comfort and implementing the protocols required to minimize the risk of RAO must be part of quality control.
* Several procedural parameters are related to the risk of RAO but hemostasis is a critical period.
* Despite the fact that non-occlusive hemostasis of the radial artery is a recognized and effective technique for reducing the risk of RAO, it is rarely practiced because it is tedious, involves additional care and is not always effective with current hemostasis systems.
* Prophylactic compression of the cubital artery during radial artery hemostasis has been shown to be effective in maintaining non-occlusive hemostasis but requires 2 devices and does not simplify care procedures.
* The Terry2™ band is a new dual device that offers effortless non-occlusive radial hemostasis and does not require repeated intervention by nursing staff.

The primary objectives of this observational study are to demonstrate the benefits, safety and impact on care of using Terry2™ band in patients undergoing diagnostic or interventional catheterization by radial (or ulnar) approach.

DETAILED DESCRIPTION:
Radial Artery Occlusion (RAO) is the most common peri-procedural complication after a trans-radial catheterization,

Although usually asymptomatic, RAO may prevent the use of radial artery access in future catheterization should the patient need one; the use And the artery cannot be used as an alternate graft in case the patient is referred for aorto-coronary bypass surgery.

Recent data has demonstrated a clinical benefit for the use of radial artery over a venous graft for patients requiring artery bypass grafts.

Current international recommendations suggest limiting the risk of RAO to less than 5% upon discharge from hospital. To do this a change of method, ie performing a non-occlusive hemostasis of the radial artery is the most effective method to limit the risk of RAO. Unfortunately, this method takes time and requires repeated interventions by nurses, which has limited its application worldwide. In addition, simple hemostasis systems (on radial artery alone) can only achieve non-occlusive hemostasis in 60-75% of cases.

On the other hand, it has been shown that by applying simultaneous pressure to the two arteries of the wrist (the radial artery and the cubital artery), one could obtain a non-occlusive hemostasis of the radial artery in more than 95% of cases and the level of RAO was reduced < 2%. However, the handling of 2 separate hemostasis systems again requires repeated intervention by the nursing staff and therefore burdens the monitoring procedure.

The device Terry2™ band applies simultaneous differential compression to the radial artery and the cubital artery. Its mechanism of action aims to accelerate the time of hemostasis, reduce nursing work, improve patient comfort and minimize the risk of radial artery occlusion during and after hemostasis.

Hypotheses:

* The Terry2™ band provides fast and safe non-occlusive radial hemostasis that limits the risk of RAO.
* The Terry2™ band is associated with increased patient comfort, reduced staff work and a minimized risk of RAO after radial catheterization.

Procedures:

At the end of the radial approach procedure, patients will have a Terry2 band installed™ according to the instructions for use. Staff will be trained on the use of the device by means of an educational video. Once the device is installed, a check for the presence of non-occlusive hemostasis will be done before the patient has returned to their room.

Once the hemostasis is completed, the permeability of the radial artery is again checked by pulse oximetry. In case of doubt about the permeability of the instrumented artery, it is recommended to validate with an ultrasound-doppler.

Rates of RAO and other access site complications, total nursing time involved and patient comfort will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for diagnostic or interventional catheterization through radial or cubital approach

Exclusion Criteria:

* Unable to understand the study design and sign an informed consent
* Unable to receive antiplatelet therapy with aspirin and/or clopidogrel-prasugrel and/or ticagrelor and intravenous anticoagulant treatment with heparin or bivalirudin
* Presence of any local conditions like hematoma or pseudo-aneurysms precluding radial or cubital access.
* Presence of PPG while simultaneously compressing the radial and cubital arteries (due to collateral branches or interosseous artery), which prevents the establishment of non-occlusive hemostasis with the Terry2(TM) band.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comer adult population referred for diagnostic or interventional catheterization by transradial or transcubital approach at the participant centers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of radial artery occlusion | 30 - 270 minutes after catheterization
  Rate of radial artery occlusion throughout hemostasis until hospital discharge as measured by oximetry (photoplethysmography PPG) .
  The absence of a PPG curve indicates radial artery occlusion. Inconclusive cases maybe confirmed by doppler echography.
Total time to hemostasis | 30 - 270 minutes after catheterization or until hemostasis is achieved
  Characterization of the total time required to obtain hemostasis of the access site after transradial catheterization using the Terry2 band.
  Measured from device installation until removal.

SECONDARY OUTCOMES:
Change in patient comfort rating | During procedure
  Change on patient comfort/pain perception measured by a visual analog scale (VAS) before placing the device and after its removal.
  The VAS used ranges from 0 to 10, where the lower scores refer to lower pain and higher comfort.
  0 -1 Very comfortable / No pain 2 -3 Comfortable / Mild pain 4 - 5 Somewhat comfortable / Moderate Pain 6 - 7 Somewhat uncomfortable / Severe Pain 8 - 9 Uncomfortable / Very severe pain 10- Very uncomfortable / Extreme pain
Rate of access site complications | up to 30 days after catheterization
  Using the EASY scale for hematoma and bleeding
Total nursing time involvement | During hemostasis up to 24 hours after catheterization.
  Total nursing time dedicated to care for access site until hemostasis is achieved. Calculated as as a combination of the number of interventions and time per intervention.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - CSSS Chicoutimi, Chicoutimi, Quebec
  - CHUM- Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Québec, Québec, Quebec
  - IUCPQ - Laval Hospital, Québec, Quebec
  - Hôpital Sainte-Marie, Trois-Rivières, Quebec